CLINICAL TRIAL: NCT00715442
Title: Phase II Non-Randomized Pre-Surgical Study Evaluating Sunitinib in Patients With Metastatic Renal Cell Carcinoma (RCC) Who Are Eligible for Cytoreductive Nephrectomy
Brief Title: Pre-Surgical Sutent in Renal Cell Carcinoma (RCC)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0511; NCI-2012-01678 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Renal Cell Carcinoma
Keywords: Kidney; Renal Cell Carcinoma; RCC; Sutent; Sunitinib malate; Clear cell; SU011248; Nephrectomy; Surgical removal of kidney; Cytoreductive nephrectomy
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib; Nephrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sunitinib + Nephrectomy (Experimental): Sunitinib 50 mg by mouth daily for 28 consecutive days. Nephrectomy will occur approximately 24 hours after the last dose of sunitinib.
  Interventions: Drug: Sunitinib; Procedure: Nephrectomy

INTERVENTIONS:
Drug: Sunitinib — 50 mg by mouth daily for 28 consecutive days
  Other Names: SU011248; Sunitinib Malate; Sutent
Procedure: Nephrectomy — Nephrectomy will occur approximately 24 hours after the last dose of sunitinib.
  Other Names: Surgical Removal of Kidney

SUMMARY:
The goal of this clinical research study is to learn if Sutent® (sunitinib malate), given before surgery, can help control renal cell carcinoma. The safety of sunitinib malate will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

Sunitinib malate is designed to block pathways that control important events such as the growth of blood vessels that are essential for the growth of cancer.

Study Treatment:

If you are found to be eligible to take part in this study, you will take sunitinib malate once a day (either with or without food) for 4 weeks in a row, followed by 2 weeks of rest with no study drug. These 6 weeks are considered 1 cycle of study treatment.

During Cycle 2, you will have surgery to remove the tumor. You will start taking sunitinib malate again after surgery (at least 14 days after surgery) on the same schedule as before.

Study Visits:

At the beginning of each new cycle (Cycles 1-6), you will have the following tests:

* Your complete medical history will be recorded.
* You will have a physical exam, including measurement of your vital signs, and weight.
* You will have a performance status evaluation.
* You will be asked about any medicines you are currently taking and if you have experienced any side effects since your last visit.
* You will have blood drawn (about 4 teaspoons) for routine testing. This blood will also be tested to check the function of your thyroid gland.
* You will have follow-up scans (the same ones you had during screening to check the disease status) at the beginning of Cycle 2, after you have surgery, and at the beginning of each of the next 4 cycles.
* You will have an ECG to measure the health of your heart.

Every 2 Cycles, you will have a follow-up echocardiogram or MUGA scan to check your heart function, if your doctor feels it is needed.

Beginning in Cycle 7, you will be asked to return to the clinic every other cycle (about every 12 weeks), unless your doctor thinks you should return more often. This means you would return for clinic visits at the start of Cycles 8, 10, 12, and so on, and may be asked to come back at other times.

At each visit, you will have the following tests:

* Your complete medical history will be recorded.
* You will have a physical exam, including measurement of your vital signs and weight.
* You will have a performance status evaluation.
* You will be asked about any medicines you are currently taking and if you have experienced any side effects since your last visit.
* You will have blood drawn (about 4 teaspoons) for routine testing at the beginning of each cycle. If you are scheduled to return to M. D. Anderson every 2 cycles (12 weeks), you may have the blood drawn for routine tests at your local doctor's office during the "non-visit" cycles.
* You will have an ECG to measure the health of your heart.
* You will have an echocardiogram or MUGA scan to check your heart function, if your doctor feels it is needed.
* You will have follow-up scans (the same ones you had during screening to check the disease status).

Length of Study:

You will continue taking sunitinib malate on this study, unless the disease gets worse, you experience intolerable side effects, and/or you need an alternative treatment during the course of the study.

Early Withdrawal:

Early withdrawal is defined as a patient not being able to complete a full cycle of sunitinib malate. If you withdraw early, you will return to clinic for the following tests:

* Your complete medical history will be recorded.
* You will have a physical exam, including measurement of your vital signs, and weight.
* You will have a performance status evaluation.
* You will have blood drawn (about 4 teaspoons) and urine collected for routine testing. This blood will also be tested to check the function of your thyroid gland.
* You will have an ECG to measure the health of your heart.
* You will be asked about any medicines you are currently taking and if you have experienced any side effects since your last visit.
* You will have follow-up scans (the same ones you had during screening to check the disease status).

Post Treatment Evaluation (within 1 month of the last dose):

About 30 days after your last dose of sunitinib malate, you will return to the clinic for a follow-up visit. You will have the following tests:

* Your complete medical history will be recorded.
* You will have a physical exam, including measurement of your vital signs, and weight.
* You will have a performance status evaluation.
* You will have blood drawn (about 4 teaspoons) and urine collected for routine testing. This blood will also be tested to check the function of your thyroid gland.
* You will be asked about any medicines you are currently taking and if you have experienced any side effects since your last visit.
* You will have follow-up scans (the same as at screening) to check the status of the disease.
* You will have an ECG to measure the health of your heart.

Long-Term Follow-Up:

Following the post-treatment visit, you will be contacted regularly to check the status of the disease. You will be contacted (by telephone or routine clinic visit) every 6-12 weeks for the first 2 years, and every 6 months after that for up to 5 years.

This is an investigational study. Sunitinib malate is commercially available and FDA approved for treatment of clear-cell renal cell carcinoma. At this time, its use in combination with surgery is for research only. Up to 50 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed metastatic clear cell RCC who are eligible for cytoreductive nephrectomy. The determination of resectability will ultimately lie in the clinical judgment of the urologist and medical oncologist involved in the care of the patient.
2. Measurable disease is defined as a lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) and measures >/= 20 mm with conventional techniques or >/= 10 mm with spiral CT scan. This does not include primary tumors, which will be removed.
3. ECOG performance status </= 1.
4. Patients must have adequate organ and marrow function within 14 days as defined below: a) absolute neutrophil count >/= 1,500/microL b) platelets >/= 75,000/microL c) Hgb > 9.0 g/dL (may be transfused or receive epoetin alfa [e.g., Epogen®] to maintain this level) d) total bilirubin </= 2.0 mg/dl • serum creatinine </= 1.5 times the upper limit of normal (ULN) e) AST(SGOT) and/or ALT (SGPT) </= 2.5 X institutional ULN for subjects without evidence of liver metastases f) AST(SGOT) and/or ALT (SGPT) </= 5 X institutional ULN for subjects with documented liver metastases
5. Female patients of childbearing potential (i.e. premenopausal, no hysterectomy) must have a normal plasma beta human chorionic gonadotropin (betaHCG) within 24 hours prior to enrolling in the study due to the possible teratogenic effect. Patients with an elevated betaHCG will undergo appropriate evaluation to rule out pregnancy (i.e. referral to Gyn service, pelvic ultrasound) and if pregnancy is ruled out and elevated betaHCG is determined to be of tumor origin, patients will be permitted to proceed on study.
6. Patients of child fathering or childbearing potential must agree to practice a form of medically acceptable birth control while on study, i.e. condoms.
7. Patients must give written informed consent prior to initiation of therapy, in keeping with the policies of the institution. Patients with a history of major psychiatric illness must be judged able to fully understand the investigational nature of the study and the risks associated with the therapy. The only approved consent is attached to this protocol.

Exclusion Criteria:

1. Patients must not have organ allografts.
2. Patients must not have had major surgical procedure, open biopsy, or significant traumatic injury within 14 days prior to Day 0, or anticipation of need for major surgical procedure during the course of the study (other than defined by protocol); or fine needle aspirations or core biopsies within 7 days prior to Day 0.
3. No prior malignancy is allowed, except for non-melanoma skin cancer, in situ carcinoma of any site, or other cancers for which the patient has been adequately treated and disease free for 2 years.
4. Patients must not have received any prior anticancer therapy for renal cell carcinoma. Radiation therapy is allowed if > 2 weeks from study drug administration.
5. Patients must not be scheduled to receive another experimental drug while on this study. Patients are permitted to be on concomitant bisphosphonates and megestrol acetate.
6. Patients must not have a primary brain tumor (excluding meningiomas other benign lesions), any brain metastases, leptomeningeal disease, seizure disorders not controlled with standard medical therapy, history of stroke within the past year.
7. History of serious systemic disease, including myocardial infarction or unstable angina within the last 12 months, history of hypertensive crisis or hypertensive encephalopathy, uncontrolled hypertension (blood pressure of > 140/90 mmHg) at the time of enrollment, New York Heart Association (NYHA) Grade II or greater congestive heart failure, unstable symptomatic arrhythmia requiring medication (subjects with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal supraventricular tachycardia are eligible), significant vascular disease or symptomatic peripheral vascular disease.
8. Patients must not have history of other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications.
9. Patients receiving any concomitant systemic therapy for renal cell cancer are excluded, but patients taking bisphosphonates and megestrol acetate are not excluded.
10. Patients must not require total parenteral nutrition with lipids.
11. Patients must not have clinical history of coagulopathy, bleeding diathesis or thrombosis within the past year.
12. Patients must not have serious, non-healing wound, ulcer, or bone fracture.
13. Pregnancy (positive pregnancy test) or lactation.
14. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment.
15. Know hypersensitivity to any component of sunitinib.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-06-24 (Actual); Primary Completion 2026-12-04 (Estimated); Study Completion 2026-12-04 (Estimated)

PRIMARY OUTCOMES:
Time to progression (TTP) | Baseline start of treatment to disease progression; up to 5 years
  TTP is defined as the time interval between treatment starts and disease progression or death, whichever occurred first, assessed each cycle (42 days).
Toxicity of Sunitinib in Patients With Metastatic Renal Cell Carcinoma (RCC) | Start of study drug up to 30 days after study drug stopped
  Toxicity defined as any Grade 3 or greater perioperative complications attributable to sunitinib.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jonasch, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Gatto F, Bratulic S, Jonasch E, Limeta A, Maccari F, Galeotti F, Volpi N, Lundstam S, Nielsen J, Stierner U. Plasma and Urine Free Glycosaminoglycans as Monitoring and Predictive Biomarkers in Metastatic Renal Cell Carcinoma: A Prospective Cohort Study. JCO Precis Oncol. 2023 Feb;7:e2200361. doi: 10.1200/PO.22.00361. PMID 36848607
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org